CLINICAL TRIAL: NCT02755428
Title: Safety and Efficacy of Subretinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigment Epitheliums in Treatment of Age-related Macular Degeneration Diseases
Brief Title: Subretinal Transplantation of Retinal Pigment Epitheliums in Treatment of Age-related Macular Degeneration Diseases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Qi Zhou, The vice President and deputy director of Institute of zoology, chinese academy of sciences, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChineseASZQ-001
Record Dates: First submitted 2016-03-26; First posted 2016-04-28 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2017-12

CONDITIONS: Dry Age-related Macular Degeneration

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- retinal pigment epithelium transplantation (Experimental): Subretinal transplantation of human embryonic stem cell derived retinal pigment epitheliums.
  Interventions: Biological: retinal pigment epithelium transplantation

INTERVENTIONS:
Biological: retinal pigment epithelium transplantation — Transplant retinal pigment epithelium derived from human embryonic stem cells into subretinal space of patients with dry age-related macular degeneration(dry AMD).

SUMMARY:
This project intends to transplant human embryonic stem cells derived retinal pigment epitheliums into subretinal space of patients to treat dry age-related macular degeneration(dry-AMD).And we will assess the safety and efficacy of RPE transplants to treat dry AMD.

DETAILED DESCRIPTION:
This project intends to transplant human embryonic stem cells derived retinal pigment epitheliums into subretinal space to treat age-related macular degeneration(AMD).

Through the statistical analysis EDTRS, BCVA, OCT, ERG, Fluorescein angiography, Ophthalmic AB ultrasound changes between before and after the treatment to assess the efficacy and safety of RPE transplants to treat AMD disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-80 years;
* Clinical diagnosis is consistent with the definition of late dry AMD in the age-related eye disease study (AREDS) (with one or more >250 micron geographic atrophy in the fovea;
* No CNV;
* The BCVA of target eye will not be better than 20/200;
* -8.00D<diopter<+8.00D，21mm<axis oculi≤28mm;
* voluntary as test subjects, signed informed consent, regular follow-up on time.

Exclusion Criteria:

* The macular atrophy caused by other diseases in addition to AMD;
* Suffer from retinitis pigmentosa, choroidal retinitis, central serous chorositis, diabetic retinopathy or other retinal vascular and degenerative diseases besides AMD;
* Lens opacities (affecting the central vision), glaucoma, uveitis, retinal detachment, optic neuropathy and other ocular history;
* Other intraocular surgery history besides cataract surgery;
* In the last 6 months, there were severe heart failure (New York Heart Association grade III and IV) or the left ventricular ejection fraction <35% in any examinations
* One of the following circumstances: (1) dialysis or eGFR<20ml/min/1.73m2; (2) urinary protein / urinary creatinine is ≥1g/g; (3) creatinine or albumin / urinary creatinine is ≥600mg/g;
* Chronic liver disease, ALT increased >3 times normal value of the upper limit;
* Combined with other serious systemic diseases, such as cor pulmonale, severe COPD (FEV1%<50%) and so on;
* Combined with severe infectious diseases (such as HIV, syphilis antibody positive, etc;
* The quantitative detection of HCV-RNA was positive, the quantitative detection of HBV-DNA was greater than 103 IU/ml, and tuberculosis was in the contagious period, etc;
* Patients who are using anticoagulant, or the platelet function is still not restored to normal after stopping antiplatelet drugs for 10 days（The results of VerifyNow test show that AUC is greater than 470 and PRU is more than 208）;
* Abnormal blood coagulation function or other obvious abnormal laboratory test results;
* Malignant tumor and history of malignant tumor;
* Women who are pregnant，prepare to be pregnant during the trial, be lactating；men who prepare to have baby during the trial;
* Any immune deficiency;
* Glucocorticoids or immunosuppressive drugs have been used in the last 3 months;
* Antipsychotic drugs have been used in the last 3 months, such as antidepressants, antipsychotic drugs, and so on;
* With hypersensitivity to tacrolimus or other macrolides;
* The history of addiction to alcoholism or prohibited drugs;
* Being participating in any intervention clinical trials;
* Poor compliance, difficult to complete the study;
* The person who did not receive the informed consent;
* Some researchers believe that there may be situations that can increase risks of the subjects or interfere clinical trials (for example, patients are prone to mental stress, depression, mental disorders, cognitive dysfunction, etc.).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
safety and tolerance of transplantation | one year
  The safety and tolerance of transplantation of clinical grade hESC-derived RPE will be considered safe: no above moderate adverse events or severe adverse events which related to transplantation of retinal pigment epithelial cells ; Cells without infectious; No tumorigenicity. Through the clinical signs of subjects and laboratory examination to judge the tolerance, integrity, repellency of RPE cells, and monitoring the presence of local or systemic infection, and presence of metastatic tumor cells.

SECONDARY OUTCOMES:
Efficacy:Early treatment of diabetic retinopathy eye chart (ETDRs) | one year
  Visual function measure: change in visual acuity
Efficacy：Best corrected visual acuity（BCVA） | one year
  Visual function measure: change in visual acuity
Efficacy：Optical coherent tomography (OCT) | one year
  Transplant and host retina integrity and survival
Efficacy：fundus autofluorescence | one year
  Transplant and host retina integrity and survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Qi, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided